CLINICAL TRIAL: NCT06034912
Title: Fundus Effects of Repeated Low-Level Red-Light Therapy in Chinese Myopic Minors: A Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Ma, Professor at Sun Yat-sen University, Chief Physician at Sun Yat-sen University Hospital, and Doctoral Supervisor at Sun Yat-sen University., Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RLRL RCT
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Red Laser Light-Induced Retinopathy of Both Eyes (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Intensity Red Light Therapy (Experimental): Intervention method：Daily wearing myopia frame glasses (optical monofocal lenses) and Low-Intensity Red Light therapy during the study to control myopia.
  Interventions: Device: Low-Intensity Red Light Therapy
- Control group (No Intervention): Intervention method: Daily wearing myopia frame glasses (optical monofocal lenses) during the study, no other treatment is used to control myopia.

INTERVENTIONS:
Device: Low-Intensity Red Light Therapy — myopia and amblyopia comprehensive treatment instrument red light feeding treatment
  Arms: Low-Intensity Red Light Therapy

SUMMARY:
1. Research Objective: The primary objective is to investigate the short-term effects of repetitive low-intensity red light therapy on the fundus of the eyes of underage individuals with myopia.
2. Research Design: This experiment employs a prospective, single-center, randomized, controlled clinical research design.
3. Primary Outcome: Changes in macular sensitivity (microperimetry).
4. Recruitment and Participant Information: The study population consists of individuals aged 7 to 17 years old. It is anticipated that there will be 35 participants in both the control group and the experimental group.
5. Trial Location: Zhongshan Ophthalmic Center, Sun Yat-sen University. Contact Information: Shuyu Chen, +190805155537, chenshuyu980916@163.com.

DETAILED DESCRIPTION:
1. Research Design: This study is an interventional research aimed at investigating the short-term effects of repeated low-intensity red light therapy on the fundus of underage individuals with myopia. Retinal light damage typically occurs in the photoreceptor layer and retinal pigment epithelium. Optical coherence tomography angiography (OCTA), OCT, pattern visual evoked potentials (VEP), microperimetry, and multifocal electroretinography (ERG) will be utilized to assess the functionality of the retina, choroid, and optic nerve, thus identifying potential areas of damage. This will provide a scientific basis for further evaluating the safety of low-intensity red light therapy.
2. Participant Recruitment:

(1) Age range: 7 to 17 years old. (2) Spherical equivalent refraction (SER): -1.00D to -5.00D. (3) Astigmatism: ≤ 2.50D. (4) Anisometropia (difference between the two equivalent spherical lenses): ≤ 1.50D.

(5) Best corrected visual acuity (BCVA) in either eye: ≥ 20/20. (6) Willingness to undergo low-intensity red light treatment. (7) Ability to comprehend the trial's purpose, voluntary participation, and signing of an informed consent form by the subject and their legal guardian.

3.Intervention:Control Group: Daily wear of frame glasses for refractive correction, without any additional treatment for myopia control.Experimental Group: Daily wear of frame glasses for refractive correction, along with low-intensity red light therapy as prescribed by the optometrist.

4.Data Collection: All examinations are conducted by experienced doctors，technicians, and optometrists during objective assessments. Data collection forms are incorporated into the medical records. Specialized research coordinators conduct regular follow-up with all subjects via telephone or WeChat.

5.Ethical Review: The trial protocol was developed before the clinical trial commenced and received approval from the ethics committee.

6.Results and Analysis: Data statistical analysis will be performed using SPSS 26.0 statistical software. The Kolmogorov-Smirnov test will be employed for normality distribution testing. Variables following a normal distribution will be expressed as mean ± standard deviation (Mean±SD). Between-group comparisons will be conducted using one-way analysis of variance. Paired t-tests will be used for pre- and post-red light exposure data. Non-normally distributed data will be expressed as median (interquartile range) [M(Q)] and analyzed using rank-sum tests. A significance level of P < 0.05 will indicate statistically significant differences.

7.Safety and Side Effects: None. 8.Discussion and Conclusion: None.

ELIGIBILITY:
Inclusion Criteria:

1. 7~17 years old；
2. Spherical equivalent refraction (SER) -1.00 to -5.00D；
3. Astigmatism≤ 2.50D；
4. Anisometropia (difference between the two equivalent spherical lenses) ≤ 1.50D；
5. Best corrected visual acuity (BCVA) in either eye ≥ 20/20；
6. Currently willing to use low-intensity red light treatment；
7. Be able to understand the purpose of the trial, voluntarily participate and have the subject and his legal guardian sign an informed consent form.

Exclusion Criteria:

1. strabismus (apparent strabismus) or amblyopia；
2. Correction of abnormal vision in either eye；
3. Any eye disease that may be related to myopia or affect refractive development, such as history of photosensitivity, macular disease, moderate to severe dry eye, corneal disease, cataract, vitreoretinal disease, infectious conjunctivitis, uveitis, optic nerve damage, congenital optic nerve development abnormalities or other eye diseases；
4. Systemic diseases, such as hypertension, lupus erythematosus, albinism, diabetes, etc；
5. previous history of convulsions, tics, central nervous system underdevelopment, psoriasis, epilepsy and psychiatric and psychological diseases；
6. used within 3 months or planned to use low-concentration atropine eye drops during the study；
7. Those who have previously used orthokeratology lenses, peripheral defocusing glasses, multifocal soft lenses and other optical therapies to control the progression of myopia, and the elution period is less than three months；
8. Other situations in which the investigator believes that the patient is not suitable to participate in this study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Latency of P1 waves | Immediately、1 day、1 month、3 months、6 months after treatment
  Multifocal electroretinogram (mfERG) was used to detect the electrophysiological activity of the local retina of the macula, and the latency of P1 wave was recorded.

SECONDARY OUTCOMES:
Amplitude and latency of P100 waves | Immediately、1 day、1 month、3 months、6 months after treatment
  Pattern visual evoked potentials (P-VEP) were used to detect the functional integrity of the visual pathway, and the amplitude and latency of the P100 wave were recorded.
Choroidal thickness | Immediately、1 day、1 month、3 months、6 months after treatment
  Optical coherence tomography (OCT) was used for choroidal thickness measurement.
Choroidal and retinal blood flow density assessment | Immediately、1 day、1 month、3 months、6 months after treatment
  Optical coherence tomography angiography (OCTA) was used to scan the choroidal and retinal scans of both eyes to check the blood flow density .
Changes in visual acuity in the macula (microperimetry) | Immediately、1 day、1 month、3 months、6 months after treatment
  All participants were treated with a microperimetry for fundus imaging and microperimetry examination without mydriasis.
Amplitude of P1 waves | Immediately、1 day、1 month、3 months、6 months after treatment
  Multifocal electroretinogram (mfERG) was used to detect the electrophysiological activity of the local retina of the macula, and the amplitude of P1 wave (expressed by reaction density) was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ma Jin, professor, Study Chair — Professor at Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Zhongshan Ophthalmic Center (Zhujiang New Town Campus), Guangzhou, China

IPD SHARING:
Plan to Share IPD: No